CLINICAL TRIAL: NCT06650865
Title: Effect of Baduanjin on Pain, Balance and Kinesiophobia in Individuals With Knee Osteoarthritis
Brief Title: Effect of Baduanjin on Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep HOŞBAY, Assoc Prof. Dr, PhD, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 145361
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional Exercise Group (Active Comparator): The routine exercise program applied to individuals with osteoarthritis who applied to the orthopedic clinic where the data will be obtained is given below.
  1st week exercises
  * Isometric quadriceps set
  * Terminal knee extension
  * Knee extension at 90 degrees flexion
  * Isometric gluteus maximus exercises
  Exercises added in week 2
  * Four-way straight leg raises
  * Bridge exercise
  * Fingertip elevation
  Exercises added in week 4
  * Mini squat (0-30 degrees)
  * Getting up from a chair without support
  * Leg press exercise with Theraband
  Exercises added in week 6
  * Stepping up and down
  * Exercises for rising on one leg
  * Semi squat (0-60 degrees)
  The exercise program will be taught to the patient and given as a home program.
  Interventions: Other: Traditional Exercise Group
- Baduanjin Exercise Group (Experimental): Standard Physical Therapy Program + Baduanjin exercises
  Baduanjin exercises An important complementary part of Qigong, the Baduanjin exercise (Eight Part Exercises or Eight Part Brocades) consists of eight different postures (supporting the chest, drawing arcs to both sides, raising one hand, practicing looking back, waving the hand and wagging the tail, touching the feet with both hands, climbing with both hands and relaxing the back).
  The exercise program will be taught to the patient and given as a home program.
  Interventions: Other: Baduanjin Exercise Group
- Telerehabilitation group (Experimental): Baduanjin exercise will be applied simultaneously with the telerehabilitation method.
  Standard Physical Therapy Program + Baduanjin exercises
  Baduanjin exercises An important complementary part of Qigong, the Baduanjin exercise (Eight Part Exercises or Eight Part Brocades) consists of eight different postures (supporting the chest, drawing arcs to both sides, raising one hand, practicing looking back, waving the hand and wagging the tail, touching the feet with both hands, climbing with both hands and relaxing the back).
  The exercise program will be taught to the patient and given as a home program.
  Interventions: Other: Telerehabilitation Group

INTERVENTIONS:
Other: Traditional Exercise Group — It is important for the therapist to organize a exercise program to provide pain control. The exercise program should be specific and clear to the patient.
  Exercises will be applied to this group. The exercise steps will be continued 3 days a week for 6 weeks. All scales and tests will be completed again at week 12 for long-term follow-up.
  Other Names: exercise
  Arms: Traditional Exercise Group
Other: Baduanjin Exercise Group — In addition to the standard physical therapy program, Baduanjin will be applied for 30 minutes.
  The exercise steps will be continued 3 days a week for 6 weeks. All scales and tests will be completed again at week 12 for long-term follow-up.
  Other Names: exercise
  Arms: Baduanjin Exercise Group
Other: Telerehabilitation Group — Baduanjin exercise will be applied simultaneously with the telerehabilitation method. In addition to the standard physical therapy program, Baduanjin will be applied for 30 minutes.
  The exercise steps will be continued 3 days a week for 6 weeks. All scales and tests will be completed again at week 12 for long-term follow-up.
  Other Names: exercise
  Arms: Telerehabilitation group

SUMMARY:
Osteoarthritis (OA) is the most common rheumatologic disease in the world, primarily resulting in progressive cartilage destruction. It is most common in the knee joint. In this study, it is aimed to determine the effect of Baduanjin to reduce kinesiobia and increase functional exercise capacity by reducing or completely eliminating balance loss and pain in patients with knee osteoarthritis and to shed light on future studies. 60 individuals between 40 and 70 years of age with osteoarthritis will be included in the study. Individuals will be randomized into three groups. In the study, Visual Analog Scale (VAS) was used to assess the severity of pain, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used to assess physical activity level, Berg Balance Scale (BDS) was used to assess balance, Tampa Kinesiophobia Scale (TKS) was used to assess kinesiophobia, Timed Up and Go Test (TUGT) and 30 Second Sit and Stand Test were used to assess functional levels. In our study, an exercise program accompanied by a physiotherapist will be applied for 12 weeks, 3 days a week. Exercise program will be applied to the first group and Baduanjin exercises will be applied to the second group in addition to the exercise program. Baduanjin exercise will be applied to the third group synchronously with the telerehabilitation method. It is thought that both techniques applied in our study may have positive effects on pain, kinesiophobia and physical function.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a long-term chronic disease in which stiffness, pain and impaired mobility occur when bones rub against each other as a result of deterioration of the cartilage in the joints. Although the disease most commonly affects the joints in the knees, hands, feet and spine, it can also be observed in the shoulder and hip joints. Clinical symptoms of OA, which is a common joint disease, include pain, joint stiffness, weakened proprioception, impaired balance and dysfunction that severely affect quality of life.

The main aim of osteoarthritis rehabilitation is to prevent functional losses by reducing pain and increasing muscle strength. Conservative treatment, pharmacologic treatment and surgical treatment are applied in osteoarthritis rehabilitation. Exercise practices, which are recommended with a high level of evidence, are the most important building blocks of conservative treatment. In individuals with knee OA, strengthening exercises, which are the leading exercise interventions, increase strength as well as power and endurance. As a result of increased muscle strength, stress on the joint is reduced, resulting in increased correct loading and stabilization. Skeletal muscles contract isometrically, concentrically and eccentrically to support the body weight against gravity and absorb shock. Eccentric strength is an integral part of lower extremity-specific activities of daily living.

When the literature is reviewed, recent studies have shown that OA patients have positive perspectives on traditional aerobic exercise. Tai Chi has been proven to reduce pain and improve physical function. Qigong, which emerged before Tai Chi, is accepted as another traditional aerobic exercise preferred by patients with knee osteoarthritis who cannot tolerate intense physical activities. An important complementary part of qigong, the Baduanjin exercise (Eight-Part Exercises or Eight-Part Brocades) consists of eight separate postures (supporting the chest, drawing arcs to both sides, raising one hand, practicing looking back, waving the hand and wagging the tail, touching the feet with both hands, climbing with both hands and relaxing the back). Baduanjin is a set of exercises, a qigong (chi kung) practice originating in China. The term "Ba Duan Jin" means "eight pieces of brocade" or "eight silk threads" in Chinese. This series of exercises involves a series of movements involving body posture, breath control and mental concentration. The main purpose of Baduanjin is to increase the circulation of energy (chi or qi), promote balance in the body, increase flexibility and improve overall health. According to traditional Chinese medicine, the free circulation of chi and its balanced distribution throughout the body is the key to a healthy life. This exercise series aims to create a physical, mental and energetic balance.

Each can have beneficial effects on different parts of the body or on specific organs. Similar to Tai Chi, Baduanjin exercise is recognized as a multicomponent therapy that combines physical, psychosocial, cognitive and spiritual components. Compared to Tai Chi, Baduanjin exercise has fewer physical and cognitive requirements, which makes it very suitable for application in patients with knee osteoarthritis in a short time. In this study, it is aimed to determine the effect of Baduanjin to reduce kinesiobia and increase functional exercise capacity by reducing or completely eliminating balance loss and pain in patients with knee osteoarthritis and to shed light on future studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with osteoarthritis of the knee,
* 40-70 years old,
* BMI <40 kg/m2,
* Grade II and Grade III OA according to the Kellgren and Lawrence radiographic classification,
* Score of 24 and above on the Standardized Mini Mental State Examination

Exclusion Criteria:

* Underwent surgery involving the lower limbs and spine,
* History of ligament injury or joint luxation involving the lower extremity,
* Diagnosed with a neurological disease affecting the lower extremities,
* Diagnosed with cardiovascular disease,
* Not receiving any other treatment in the last 3 months
* Taking anxiolytic and sedative drugs,
* Psychiatric illness,

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain on the Visual Analog Scale (VAS) at week 12. Change from baseline in balance on the Berg Balance Scale (BDS) at week 12. | 12 weeks
  The Visual Analog Scale is a one-dimensional scale commonly used to measure pain intensity. The VAS is a 0-10 cm (0-100 mm) long measuring instrument. The scale starts with "no pain" and ends with "unbearable pain".
Change from baseline on the Western Ontario and McMaster Universities Arthritis Index (WOMAC) at week 12 | 12 weeks
  WOMAC assesses patients' pain, stiffness and physical function in the last 48 hours. A higher score indicates an increase in pain, stiffness and lack of physical function.
Change from baseline in pain on the Berg Balance Scale at week 12 | 12 weeks
  The Berg Balance Scale (BBS) is a scale that includes 14 instructions and for each instruction, the patient's performance is observed and a score between 0 and 4 is given. A score of 0 is given when the patient cannot perform the activity at all, while a score of 4 is given when the patient completes the activity independently.
Change from baseline in pain on the Timed Up & Go (TUG) Test at week 12 | 12 weeks
  The Timed Up and Go (TUG) test is a test used to determine dynamic balance and fall risk. The time it takes for a person to get up from a chair, walk three meters, turn 180 degrees, walk back to the chair and sit down while turning 180 degrees is calculated.
Change from baseline in pain on the 30-second Sit-Rise Test at week 12 | 12 weeks
  30-second Sit-Rise test is a test used to measure leg strength and endurance for 30 s.
Change from baseline in pain on the Tampa Scale of Kinesiophobia (TSK) at week 12 | 12 weeks
  The Tampa Kinesiophobia scale is a scale to measure patients' avoidance of exercise and fear of movement. A high score on the scale indicates a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brosseau L, Taki J, Desjardins B, Thevenot O, Fransen M, Wells GA, Mizusaki Imoto A, Toupin-April K, Westby M, Alvarez Gallardo IC, Gifford W, Laferriere L, Rahman P, Loew L, De Angelis G, Cavallo S, Shallwani SM, Aburub A, Bennell KL, Van der Esch M, Simic M, McConnell S, Harmer A, Kenny GP, Paterson G, Regnaux JP, Lefevre-Colau MM, McLean L. The Ottawa panel clinical practice guidelines for the management of knee osteoarthritis. Part two: strengthening exercise programs. Clin Rehabil. 2017 May;31(5):596-611. doi: 10.1177/0269215517691084. Epub 2017 Feb 1. PMID 28183213
- [Background] Dore AL, Golightly YM, Mercer VS, Shi XA, Renner JB, Jordan JM, Nelson AE. Lower-extremity osteoarthritis and the risk of falls in a community-based longitudinal study of adults with and without osteoarthritis. Arthritis Care Res (Hoboken). 2015 May;67(5):633-9. doi: 10.1002/acr.22499. PMID 25331686
- [Background] Ghandali E, Moghadam ST, Hadian MR, Olyaei G, Jalaie S, Sajjadi E. The effect of Tai Chi exercises on postural stability and control in older patients with knee osteoarthritis. J Bodyw Mov Ther. 2017 Jul;21(3):594-598. doi: 10.1016/j.jbmt.2016.09.001. Epub 2016 Sep 10. PMID 28750970
- [Background] Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC Musculoskelet Disord. 2005 Jan 28;6:3. doi: 10.1186/1471-2474-6-3. PMID 15679884
- [Background] Levinger P, Dunn J, Bifera N, Butson M, Elias G, Hill KD. High-speed resistance training and balance training for people with knee osteoarthritis to reduce falls risk: study protocol for a pilot randomized controlled trial. Trials. 2017 Aug 18;18(1):384. doi: 10.1186/s13063-017-2129-7. PMID 28821271
- [Background] Li D, Li S, Chen Q, Xie X. The Prevalence of Symptomatic Knee Osteoarthritis in Relation to Age, Sex, Area, Region, and Body Mass Index in China: A Systematic Review and Meta-Analysis. Front Med (Lausanne). 2020 Jul 16;7:304. doi: 10.3389/fmed.2020.00304. eCollection 2020. PMID 32766258
- [Background] Lockhart C, Scott BR, Thoseby B, Dascombe BJ. Acute Effects of Interset Rest Duration on Physiological and Perceptual Responses to Resistance Exercise in Hypoxia. J Strength Cond Res. 2020 Aug;34(8):2241-2249. doi: 10.1519/JSC.0000000000002755. PMID 30063554
- [Background] Xiong X, Wang P, Li S, Zhang Y, Li X. Effect of Baduanjin exercise for hypertension: a systematic review and meta-analysis of randomized controlled trials. Maturitas. 2015 Apr;80(4):370-8. doi: 10.1016/j.maturitas.2015.01.002. Epub 2015 Jan 9. PMID 25636242